CLINICAL TRIAL: NCT05474547
Title: Effect of Meditation on the Young Mental Health - A Feasibility Pilot Quasi-experimental Study
Brief Title: Meditation and Youth Mental Health
Acronym: Med-YMH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Habib University (Other)
Responsible Party: Principal Investigator, Humaira Jamshed, Assistant Professor, Habib University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HabibU
Record Dates: First submitted 2022-07-23; First posted 2022-07-26 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Healthy
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meditation (Experimental): Meditation for 30 min 10 days
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Meditation — Students will meditate for 30 min every day for 10 days

SUMMARY:
Youth is a crucial time of life when physical and mental well-being is critical. Students are vulnerable due to academic and pandemic stresses. Meditation research has been showing effects on improved parameters of mental health (sleep quality, attention, memory, and concentration), emotional wellbeing (reduced stress and anxiety), and physiological parameters (better metabolism, circulation, immunity, etc.), which influence the life and academic performance of students. This study is designed to examine the feasibility of conducting a meditation intervention among students of a small liberal arts university in Pakistan. Future larger and longer randomized controlled clinical trials on high-risk youth may be planned at a later stage to see the impact on academic performance and career progression.

ELIGIBILITY:
Inclusion Criteria:

* Healthy students

Exclusion Criteria:

* Students suffering from a serious illness
* Students already meditating regularly

Ages: 16 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-07-25 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Meditation Practice | 10 days
  Determinants of Meditation Practice Inventory
Sleep quality (sleep duration, deep sleep, light sleep, REM) | 10 days
  Sleep quality as measure by the fitness watch

SECONDARY OUTCOMES:
Physical activity and Heart Rate | 10 days
  Physical activity as measure by the the fitness watch
Stress and Breathing Score | 10 days
  Stress levels as measure by the the fitness watch
Food intake and nutrient profile | 10 days
  Dietary pattern measured through an online app

OTHER OUTCOMES:
Emotional wellbeing | 10 days
  Mental Health Continuum - Short Form MHC-SF; Each of the 14 items on the MHC-SF can be scored between 0 and 5, which means that the total score on the scale can range from 0 to 70 points. Higher scores indicate a higher level of emotional wellbeing.
Depression Anxiety and Stress | 10 days
  Depression, Anxiety and Stress Score (DASS-21); The total score on the scale can range from 0 to 21 points. Higher scores indicate Severe depression while lower score indicates mild anxiety.
Resilience and Resilience Coping | 10 days
  Brief Resilience Scale (BRS) and Brief Resilience Coping Scale (BRCS); The possible score range on the BRS is from 1 (low resilience) to 5 (high resilience). The possible score range on the BRCS is from 4 (low resilience) to 20 (high resilience).
Grit | 10 days
  Short grit scale (Grit-S). Scores can vary from 1 point (low grit) to maximally 5 points (high grit).
Loneliness | 10 days
  UP LAS; The score can range from 25 (low) to 100 (high).
Gratitude, Resentment and Appreciation | 10 days
  GRAT-Short Form; higher scores are better
Happiness | 10 days
  Oxford Happiness Questionnaire; higher score is more happiness.
Empathy | 10 days
  Empathy Quotient, This score is on a range from 0 (low level of empathy) to 80 (high level of empathy)
Internet Use | 10 days
  Generalized Problematic Internet Use Scale - GPIUS
Nomophobia Questionnaire | 10 days
  NMPQ
Social Networking Addiction | 10 days
  SNAS

CONTACTS AND LOCATIONS:
Overall Officials: Humaira Jamshed, PhD, Principal Investigator — Integrated Sciences and Mathematics, Dhanani School of Science and Engineering, Habib University

IPD SHARING:
Plan to Share IPD: No